CLINICAL TRIAL: NCT03490942
Title: Fixed Rate Continuous Subcutaneous Glucagon Infusion (CSGI) vs Placebo in Type 1 Diabetes Mellitus Patients With Recurrent Severe Hypoglycemia: Effects on Counter-Regulatory Responses to Insulin-Induced Hypoglycemia
Brief Title: Glucagon Infusion in T1D Patients With Recurrent Severe Hypoglycemia: Effects on Counter-Regulatory Responses
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Primary endpoint was not met
Sponsor: Xeris Pharmaceuticals (Industry)
Collaborators: Integrated Medical Development (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: XSGO-AF01
Record Dates: First submitted 2018-03-25; First posted 2018-04-06 (Actual); Results first posted 2021-02-21 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2020-05

CONDITIONS: Hypoglycemia Unawareness; Diabetes Mellitus, Type 1
Keywords: glucagon; hypoglycemia counter-regulation
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Glucagon

STUDY DESIGN:
Intervention Model Description: This is a prospective, randomized, controlled, double-blind, parallel 4-group trial with the primary analysis after 4 weeks treatment with CSGI or placebo.
Who Masked: Participant, Investigator
Masking Description: double-blind, placebo-controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- CSGI high infusion rate (Experimental): Glucagon given as a continuous subcutaneous infusion for 28 days
  Interventions: Drug: Glucagon
- CSGI low infusion rate (Experimental): Glucagon given as a continuous subcutaneous infusion for 28 days
  Interventions: Drug: Glucagon
- Placebo high infusion rate (Placebo Comparator): Placebo given as a continuous subcutaneous infusion for 28 days
  Interventions: Drug: Placebo
- Placebo low infusion rate (Placebo Comparator): Placebo given as a continuous subcutaneous infusion for 28 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Glucagon — CSI-Glucagon is a room temperature stable, non-aqueous, liquid formulation of glucagon.
  Other Names: CSI-Glucagon; CGSI
  Arms: CSGI high infusion rate; CSGI low infusion rate
Drug: Placebo — The placebo solution is a non-active formulation containing excipients only.
  Arms: Placebo high infusion rate; Placebo low infusion rate

SUMMARY:
This is a prospective, randomized, controlled, double-blind, parallel 4-group trial with the primary analysis after 4 weeks of treatment with continuous subcutaneous glucagon infusion (CSGI) or placebo. After a 1-week qualification on continuous glucose monitoring (CGM), subjects will have their baseline hypoglycemia counter-regulatory response hormones quantified using a step-wise hypoglycemia induction procedure. Subjects meeting eligibility requirements will be randomized to 1 of 4 treatment groups, 2 glucagon, 2 placebo. Subjects will receive blinded study drug for 4 weeks, and they will be followed for an additional 26 weeks post-treatment. Subjects' counter-regulatory hormone response will be measured at baseline, the end of treatment (4 weeks), and 13 and 26 weeks after treatment ends.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females diagnosed with type 1 diabetes mellitus for at least 24 months.
2. Random serum C-peptide concentration < 0.5 ng/ml at Screening.
3. Current use of multiple daily dosing insulin treatment < 1 U/(kg*day) total daily dose either administered with subcutaneous injections or continuous subcutaneous insulin infusion (CSII).
4. Recurrent severe hypoglycemia as defined by minimally two events during the last year and at least one the last six months requiring not merely receiving third party intervention and either confirmation with a measured glucose < 50 mg/dl, or prompt recovery from impaired consciousness. Events must be documented in patient chart prior to study entry. Events induced as a part of clinical diagnostics or experimentation do not qualify.
5. Performs monitoring of glucose minimally 3 times a day. Patients using continuous glucose monitoring for monitoring should continue to do so during the course of the study.
6. Age 21-64 years, inclusive, at screening.
7. Willingness to provide informed consent and follow all study procedures, including using the Medtronic smart phone application "iPRO2mylog" for diabetes data logging and attending all scheduled visits.

Exclusion Criteria:

1. Subjects using CSII, who do not use a Medtronic pump.
2. Hemoglobin A1c ≥9.0% at Screening.
3. Chronic kidney disease stage 4 or 5.
4. Hepatic disease, including serum alanine transaminase (ALT) or aspartate transaminase (AST) greater than or equal to 3 times the upper limit of normal; hepatic synthetic insufficiency as defined as serum albumin < 3.0 g/dL; or serum bilirubin > 2.0.
5. Hematocrit of less than or equal to 30% at Screening.
6. Blood pressure (BP) reading at Screening where systolic BP <90 or >150 mm Hg, or diastolic BP <50 or >100 mm Hg.
7. Clinically significant echocardiogram (ECG) abnormalities at Screening.
8. Congestive heart failure, New York Heart Association (NYHA) class II, III or IV,
9. History of myocardial infarction, unstable angina or revascularization within the past 6 months.
10. History of a cerebrovascular accident.
11. Current seizure disorder.
12. History of pheochromocytoma or disorder with increased risk of pheochromocytoma (multiple endocrine neoplasia type 2, neurofibromatosis, or Von Hippel-Lindau disease).
13. History of insulinoma.
14. Active malignancy within 5 years from Screening, except basal cell or squamous cell skin cancers. History of breast cancer or malignant melanoma will be exclusionary.
15. Major surgical operation within 30 days prior to Screening.
16. Current bleeding disorder, treatment with warfarin, or platelet count below 50,000 at Screening.
17. History of allergies to glucagon or glucagon-like products, or any history of significant hypersensitivity to glucagon or any related products or to any of the excipients in the investigational formulation.
18. History of glycogen storage disease.
19. Any concurrent illness, other than diabetes, that is not controlled by a stable therapeutic regimen.
20. Whole blood donation of 1 pint (500 mL) within 8 weeks prior to Screening. Donations of plasma, packed red blood cells, platelets or quantities less than 500 mL are allowed at investigator discretion.
21. Active substance or alcohol abuse (more than 21 drinks/wk. for males or 14 drinks/wk. for females). Subjects reporting active marijuana use and/or testing positive for tetrahydrocannabinol via rapid urine test will be allowed to participate in the study at the discretion of the investigator. Subjects positive for other drugs of abuse via rapid urine test who report use of a prescription or over-the-counter medication that would explain such a finding will be allowed to participate at the discretion of the investigator.
22. Administration of glucagon within 14 days of Screening.
23. Pregnant and/or Lactating. For subjects of childbearing potential, there is a requirement for a negative urine pregnancy test and for agreement to use contraception and to refrain from breast feeding during the study and for at least 1 month after participating in the study. Acceptable contraception includes birth control pill / patch / vaginal ring, Depo-Provera, Norplant, an intra-uterine device, the double barrier method (the female uses a diaphragm and spermicide and the male uses a condom), or abstinence.
24. Inadequate venous access.
25. Participation in other studies involving administration of an investigational drug or interventional device within 30 days or 5 half-lives, whichever is longer, before Screening for the current study and during the four weeks of study product administration in the current study.
26. Any reason the principal investigator deems exclusionary.

Ages: 21 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2018-03-15 (Actual); Primary Completion 2019-11-04 (Actual); Study Completion 2020-02-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - University of Alabama, Birmingham, Birmingham, Alabama
  - University of California, San Diego, San Diego, California
  - Emory University - Grady Memorial Hospital, Atlanta, Georgia
  - Atlanta Diabetes Associates, Atlanta, Georgia
  - University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CSGI High Infusion Rate | CSGI Low Infusion Rate | Placebo High Infusion Rate
Started | 15 | 18 | 16
Completed | 5 | 8 | 9
Not Completed | 10 | 10 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CSGI High Infusion Rate | CSGI Low Infusion Rate | Placebo High Infusion Rate | Total
Number analyzed (Participants) | 15 | 17 | 16 | 48
Age, Continuous [Median (Full Range); unit: years] | 47 [27 to 61] | 37 [22 to 60] | 39 [21 to 61] | 41.5 [21 to 61]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 11 | 8 | 29
  Male | 5 | 6 | 8 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 4 | 0 | 5
  Not Hispanic or Latino | 14 | 13 | 16 | 43
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 4 | 3 | 2 | 9
  White | 11 | 13 | 13 | 37
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Plasma Epinephrine
Description: Plasma epinephrine concentration after 30 minutes of induced hypoglycemia. Change from baseline to the end of treatment will be assessed.
Time Frame: 0-30 minutes
Measure: Mean (Standard Deviation); unit: Pg/mL
Arm/Group | CSGI High Infusion Rate | CSGI Low Infusion Rate | Placebo High Infusion Rate
Number analyzed (Participants) | 14 | 17 | 14
Pg/mL | 100.0 (150.10) | 144.4 (168.56) | 167.3 (138.87)

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | CSGI High Infusion Rate | CSGI Low Infusion Rate | Placebo High Infusion Rate
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/17 | 0/16
Serious Adverse Events (participants affected / at risk) | 2/15 | 0/17 | 0/16
Other Adverse Events (participants affected / at risk) | 7/15 | 4/17 | 2/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CSGI High Infusion Rate (N=15) | CSGI Low Infusion Rate (N=17) | Placebo High Infusion Rate (N=16)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | NA | NA — Subject 03-04, a 31-year-old male in the high rate CSGI group, had a treatment-emergent SAE of foot fracture on Study Day 102, as a result of an accident with a chainsaw.
Gastric emptying (Gastrointestinal disorders) | 1 (1) | NA | NA — SAE of impaired gastric emptying on Study Day 100. This subject had a medical history of gastroparesis. The SAE was moderate in intensity, did not result in study discontinuation, was considered not related to study drug by the Investigator
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CSGI High Infusion Rate (N=15) | CSGI Low Infusion Rate (N=17) | Placebo High Infusion Rate (N=16)
Nausea (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 (0) — Nausea
Vomiting (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0) — Vomiting
Headache (General disorders) | 2 (2) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) — Redness of the skin

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-12-21): https://cdn.clinicaltrials.gov/large-docs/42/NCT03490942/Prot_000.pdf
  • Statistical Analysis Plan (2019-12-21): https://cdn.clinicaltrials.gov/large-docs/42/NCT03490942/SAP_001.pdf